CLINICAL TRIAL: NCT03776344
Title: Efficacy of Virtual Reality for Post Operative Pain: A Randomized Controlled Trial
Brief Title: Virtual Reality for Post Operative Pain
Acronym: VRppain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Raluca Georgescu, Phd student, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7150
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: We tested the efficacy of a VR environment in the treatment of pain after surgery.
Who Masked: Participant, Care Provider
Masking Description: As we had two groups in which one used a device for ensuring the masking the entire procedure was conducted in a separate room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Patients randomized to the experimental group will benefit from the usual standard care following surgery and during the second day the opportunity to use virtual reality for 15 minute. Along VR, they will complete the psychological and physiological measures.
  Interventions: Device: Virtual Reality intervention - Oculus Rift HD
- Non-VR condition (Standard of Care) (No Intervention): Patients randomized to the control group will benefit from the usual standard care following surgery and during the second day will complete the psychological and physiological measures.

INTERVENTIONS:
Device: Virtual Reality intervention - Oculus Rift HD — During the VR experience patients will have the opportunity to choose from different VR environments (VR application - Nature Treks VR) and explore them using Oculus Rift Device.
  Arms: Virtual Reality

SUMMARY:
Randomized controlled trial to measure pain experience, side effects and satisfaction of VR following varicose vein, hernia repair and gallbladder surgeries.

DETAILED DESCRIPTION:
While there is substantial evidence supporting the use of Virtual Reality (VR) during dressing changes for burn victims, there are little information of the effect of VR to decrease pain after surgery. Although pharmacological analgesics are popular in clinical practice, this approach usually is associated with side effects, most commonly nausea, cognitive dysfunction, and constipation. Generally, VR effects are based on gate theory of cognitive load, due to the fact that conscious attention is needed to perceive pain and we can process a finite amount of information.High-Tech-VR devices shown to be more effective in reducing pain than are Low-Tech-VR systems (Prothero, J. D., & Hoffman, H. D, 1995). In addition, studies have shown that interactivity play an important role to decrease both, pain unpleasantness and time spent thinking about pain, while increasing fun (Wender, R., et al., 2010, Gromala, D., et al 2011). Thus, interactivity helps patients to have a better immersion into VR world. Considering this, in the proposed study, patients will be randomized to either receive a high immersive and interactive VR environment using Oculus Rift Headset in addition to standard care or to receive only standard care during their post-operative care following surgery to prospectively assess the utility of virtual reality (VR) for pain management following varicose vein, hernia repair and gallbladder surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient with varicose vein, hernia repair or gallbladder surgery
* Patient in the acute care units, 1-3 days following surgery.
* Willing and able to provide informed consent and participate in the study visit and study follow-up questionnaire.

Exclusion Criteria:

* Non-Romanian speaking patients.
* Age > 18 years and < 65 years.
* Patients with neoplastic pathologies.
* Patients with history of motion sickness.
* Patients with visual impairment.
* Patients with severe/profound cognitive impairments measured with Six-item Cognitive Impairment Test (6CIT).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Pain intensity before intervention; Change from Baseline pain intensity (immediately following intervention)
  Graphic Rating Scale measure pain intensity from 1 to 10, 1 - no pain; 10 - worst pain.
Pain intensity | 5 minutes before intervention (baseline)
  Skin conductance response
Pain intensity | 15 minutes - During the intervention
  Skin conductance response

SECONDARY OUTCOMES:
Satisfaction with the intervention | Immediately following intervention
  Patient Satisfaction Survey
Presence in the VR environment | Immediately following intervention
  Presence Inventory assesses the degree of spatial presence, involvement, ecological validity, overall presence, and negative effects experienced during the VR intervention
Simulator Sickness | Immediately following intervention
  Simulator Sickness Questionnaire
Relaxation | Relaxation level before intervention; Change from Baseline relaxation level (immediately following intervention)
  Graphic Rating Scale measure relaxation from 1 to 10, 1 - stressed; 10 - very relaxed.
Time thinking about pain | immediately following intervention
  Graphic Rating Scale measure the time spent thinking about pain from 1 to 10; 1 - not at all, 10 - all the time

CONTACTS AND LOCATIONS:
Locations (1):
- Municipal Hospital of Cluj-Napoca, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
All collected data will be shared in an anonymized manner.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the manuscript will be published.